CLINICAL TRIAL: NCT04964609
Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Brief Title: EmbracePlus SpO2 Accuracy Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Empatica, Inc. (Industry)
Collaborators: Empatica Srl (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-4; EMPA01 (Other: UCSF)
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Oximetry
Keywords: Oximetry; Wearable; SpO2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): Comparison of EmbracePlus SpO2 readings with arterial blood saturation laboratory analysis in the same subject
  Interventions: Device: EmbracePlus

INTERVENTIONS:
Device: EmbracePlus — A device intended for use by researchers and healthcare professionals for continuous collection of physiological parameters in home and healthcare settings.
  Parallel blood gas analysis to determine oxyhemoglobin saturation (SaO2) using an ABL-90 multi-wavelength oximeter.

SUMMARY:
The aim of this study is to test the accuracy of EmbracePlus computed SpO2 during mild, moderate and severe hypoxia (a lower-than-normal concentration of oxygen in arterial blood); ie, a range of arterial HbO2 saturations from 100 to down to 70%. This is done by comparing the reading of the the subject device during brief, steady state hypoxia with a gold-standard measurement of blood oxyhemoglobin (hemoglobin carrying oxygen) saturation, that is arterial blood sample processed in a laboratory.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, aged ≥18 and <50.
* The subject is in good general health with no evidence of any medical problems.
* The subject is fluent in both written and spoken English.
* The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

* The subject is obese (BMI>30).
* The subject has a known history of heart disease, lung disease, kidney or liver disease.
* Diagnosis of asthma, sleep apnea, or use of CPAP.
* Subject has diabetes.
* Subject has a clotting disorder.
* The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
* The subject has any other serious systemic illness.
* The subject is a current smoker.
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
* The subject has a history of fainting or vasovagal response.
* The subject has a history of sensitivity to local anesthesia.
* The subject has a diagnosis of Raynaud's disease.
* The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
* The subject is pregnant, lactating or trying to get pregnant.
* The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
* The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
SpO2 Accuracy | Through study completion, 3 months average
  SpO2 as measured by the subject device during periods of low motion will be compared to the oxyhemoglobin saturation (SaO2) as measured by direct oximetry with a Radiometer ABL-90 multi-wavelength oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- Hypoxia Research Laboratory Department of Anesthesia and Perioperative Care University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerboni G, Comunale G, Chen W, Lever Taylor J, Migliorini M, Picard R, Cruz M, Regalia G. Prospective clinical validation of the Empatica EmbracePlus wristband as a reflective pulse oximeter. Front Digit Health. 2023 Dec 4;5:1258915. doi: 10.3389/fdgth.2023.1258915. eCollection 2023. PMID 38111608